CLINICAL TRIAL: NCT06167161
Title: Clinical Investigation and Validation of a Self-fitted Air-conduction Hearing Aid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Concha Inc. (Industry)
Collaborators: University of Minnesota (Other); San Jose State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PROT-001
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Hearing Loss
Keywords: air-conduction hearing aid; over-the-counter; self-fitting
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Intervention Model Description: This investigation will incorporate a within-subject, randomized, crossover study design in which all study participants will complete two different study arm conditions. During the first visit, subjects will be randomly allocated to study arm A (clinician-fitting) or study arm B (self-fitting). Following the initial two-week take-home field trial, the research participants will be assigned to the opposite study arm such that a complete two-sequence crossover design (AB/BA design) will be followed. The same within-subject crossover design will be followed in both clinical sites and for all individuals who will be enrolled in the study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Screening, intake and first fit (either clinician-fitting or self-fitting ) (Active Comparator): This clinical trial compares two methods of fitting individuals who suffer from hearing loss with a hearing aid device. Subjects will wear the hearing aid after receiving the clinician-fitting (device fitted by a clinician according to standard clinical best practice procedures) and self-fitting (device fitted by the user directly without assistance from a clinician following an automated assessment and fitting process) for two weeks each, totaling to approximately 1 month of wear throughout the trial. During the first visit, all individuals will go through intake procedures and a basic audiologic evaluation. After this is completed, individuals will be randomly assigned into one of two arms of the study. Individuals in the first visit of the study, will receive either the clinician-fitting or the self-fitting method for the first two weeks, then will switch to the experimental self-fitting or the clinician-fitting method for the last half. The order of the fitting will be randomized.
  Interventions: Device: Hearing aid
- Second fit (either clinician-fitting or self-fitting ) (Sham Comparator): In the second visit of the study, individuals who randomly received the conventional clinician-fitting for the first two weeks (first period) will switch to the experimental self-fitting for the remainder of the study (second period). Conversely, individuals who received the experimental self-fitting method for the first two weeks (first period) will switch to the clinician-fitting method for the last two weeks (second period). The same within-subject crossover design will be followed in both clinical sites and for all individuals who were enrolled in the study.
  Interventions: Device: Hearing aid

INTERVENTIONS:
Device: Hearing aid — The hearing aid is a receiver-in-canal style hearing aid which can be programmed and adjusted by proprietary software and through a dedicated smartphone application

SUMMARY:
Approximately 48 million people in the United States have hearing loss or hearing difficulties in noisy environments. Concha Inc. is working on introducing a wireless air-conduction hearing aid to the market, featuring a self-fitting feature. Self-fitting hearing aids have emerged in recent years as a potentially viable option towards addressing unmet hearing health care needs for millions of individuals who suffer from mild-to-moderate hearing loss. The purpose of this study is to evaluate the efficiency and reliability of the self-fitting strategy developed by Concha Inc.

DETAILED DESCRIPTION:
The clinical study will be carried out using a within-subject, randomized, crossover study design in which all study participants will complete two different study arm conditions (clinician-fitting and self-fitting). Objective, subjective, and behavioral responses will be gathered from a variety of hearing-related surveys and tests, and will be analyzed quantitatively to evaluate the efficiency and reliability of the self-fitting procedure developed by Concha Inc.

The Quick Speech-in-Noise (QuickSIN) Test will be used as the primary effectiveness endpoint. QuickSIN is a quick and easy test that can measure an individual's ability to understand speech in noise. The secondary effectiveness endpoint will be assessed by using the Abbreviated Profile of Hearing Aid Benefit (APHAB). The APHAB was designed to evaluate the effect of hearing impairment or benefit in daily life APHAB and has long been considered the gold standard for patient-reported perceived benefit.

For this clinical study to be deemed successful, the self-fitting method needs to yield outcomes (namely QuickSIN and APHAB scores) which are non-inferior to the clinician-fitting method. Non-inferiority refers to an outcome where the new intervention (in our case, self-fitting) is not significantly worse than the established intervention (in our case, clinician-fitting), while also accounting for a clinically-significant margin.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18 years of age or older
* Apple iPhone X or newer (iOS 14 compatible or greater)
* Mix of male and female subjects
* Willing and able to perform all tests required for the study
* Signed and dated informed consent before the start of any study specific procedure
* Able to read and comprehend English
* Mild-to-moderate bilateral sensorineural hearing loss (defined according to thresholds from 250-8000 Hz with at least one threshold greater than 20 dB HL and thresholds at 500, 1000, 2000 and 4000 Hz less than or equal to 55, 65, 70, and 80 dB HL, respectively)

Exclusion Criteria:

* Hearing outside of limits noted, above
* Visible deformities of the ear since birth or from injury
* Fluid, pus, or blood coming out of the ear within the previous six months
* Sudden, quickly worsening, or fluctuating hearing loss within the previous six months
* Dizziness or periodic vertigo associated with hearing loss
* Hearing loss in only one ear or a large difference in hearing between ears
* Ear wax build up or feeling that something is in the ear canal
* Pain or discomfort in the ear
* Inability to follow the procedures of the study due to language problems, or other cognitive problems
* Any other history of chronic middle and outer ear disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
QuickSIN | 15 days
  A standardized measure of speech communication in noise, Quick Speech-in-Noise. (QuickSIN). Scores are clinically reported as SNR loss, the difference (in dB) between a listener's performance and that of normal-hearing adult controls. The SNR loss score is an indication of an individual's overall degree of difficulty understanding speech in noise. The greater the SNR loss the poorer the listener's ability is to hear in noise. The QuickSIN test manual provides adjective descriptors corresponding to the SNR loss score where an SNR loss score of 0 to 2 dB is normal, 2 to 7 dB is mild, 7 to 15 dB is moderate, and greater than 15 dB is defined as severe.

SECONDARY OUTCOMES:
APHAB | 15 days
  Self-report scale according to the Abbreviated Profile of Hearing Aid Benefit (APHAB). The APHAB is a self-report scale consisting of 24 Likert scale questions and is composed of four subscales including Ease of Communication (EC), Reverberation (RV), Background Noise (BN), and Aversiveness (AV). This outcome measure assesses residual activity limitations for hearing impaired individuals and it ranges from Never (1%) to Always (99%). APHAB scores represent how frequently clients experience performance problems and therefore a high APHAB score reflects a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Peggy Nelson, PhD, Principal Investigator — University of Minnesota; Anusha Yellamsetty, PhD, Principal Investigator — San Jose State University
Locations (2):
- United States (2):
  - San Jose State University, San Jose, California
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No